CLINICAL TRIAL: NCT04427072
Title: A Phase III, Randomized, Controlled, Open-label, Multicenter, Global Study of Capmatinib Versus SoC Docetaxel Chemotherapy in Previously Treated Patients With EGFR wt, ALK Negative, Locally Advanced or Metastatic (Stage IIIB/IIIC or IV) NSCLC Harboring MET Exon 14 Skipping Mutation (METΔex14).
Brief Title: Study of Capmatinib Efficacy in Comparison With Docetaxel in Previously Treated Participants With Non-small Cell Lung Cancer Harboring MET Exon 14 Skipping Mutation
Acronym: GeoMETry-III
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision not related to any safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2301; 2020-001578-31 (EudraCT Number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non small cell lung cancer; Non small cell lung carcinoma; NSCLC; INC280; capmatinib; MET mutation; MET exon14; MET exon14 skipping; MET exon14 deletion; METex14; METex14del; MET∆ex14; EGFRwt; Epidermal growth factor receptor wild type; ALK negative; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib; Docetaxel

STUDY DESIGN:
Intervention Model Description: Participants randomized to docetaxel treatment will be eligible to crossover to receive capmatinib treatment after blinded independent review committee (BIRC)-confirmed, RECIST 1.1- defined disease progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capmatinib (Experimental): 400 mg, capmatinib tablets, administered orally twice daily
  Interventions: Drug: Capmatinib
- Docetaxel (Active Comparator): Docetaxel 75 mg/m^2 solution administered by intravenous infusion on Day 1 of every 21-day cycle
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Capmatinib — 400 mg, capmatinib tablets, administered orally twice daily
  Other Names: INC280
  Arms: Capmatinib
Drug: Docetaxel — Docetaxel 75 mg/m^2 by intravenous infusion every 21 days
  Arms: Docetaxel

SUMMARY:
The purpose of the study was to learn whether the study drug (capmatinib) helps to control lung cancer better compared to a single agent chemotherapy (docetaxel) and whether it is safe when given to patients suffering from a particular type of lung cancer. This type of cancer is called non-small cell lung cancer (NSCLC) with certain specific genetic alterations (called mutations) of a gene called MET, within a specific part of the gene called exon 14.

DETAILED DESCRIPTION:
Twenty-two patients with advanced or metastatic lung cancer, with these specific mutations in the MET gene but without changes in their epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genes, were enrolled in this study. Participants were randomly assigned to get either capmatinib or docetaxel in a 2 to 1 ratio. The randomization was stratified by prior lines of systemic therapy received for advanced/metastatic disease (one line vs. two lines).

During treatment, visits were scheduled every 21 days.

For all participants, the respective treatment (either with capmatinib or docetaxel) could be continued beyond initial disease progression as per RECIST 1.1 (as assessed by the investigator and confirmed by BIRC) if, in the judgment of the investigator, there was evidence of clinical benefit, and the participant wished to continue on the study treatment. After treatment discontinuation, all participants were followed for safety evaluations during the safety follow-up period, and the participant's status was collected every 12 weeks as part of the survival follow-up.

Participants randomized to docetaxel treatment were eligible to cross over to receive capmatinib treatment after BIRC-confirmed, RECIST 1.1-defined progressive disease and after meeting the eligibility criteria prior to crossover. This was the extension treatment phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Stage IIIB/IIIC (not amenable to surgery, radiation or multi modality therapy) or IV NSCLC (according to Version 8 of the American Joint Committee on Cancer (AJCC) Staging Manual) at the time of study entry.
* Histologically or cytologically confirmed diagnosis of NSCLC that was:

  1. EGFR wt. Assessed as part of participant's standard of care by a validated test for EGFR mutations as per local guidelines. The EGFR wt status (for EGFR mutations that predict sensitivity to EGFR therapy, including, but not limited to exon 19 deletions and exon 21 L858R substitution mutations.
  2. AND ALK rearrangement negative. Assessed as part of participant's standard of care by a validated test.
  3. AND had METΔex14 mutation as determined by Novartis-designated central laboratory or by locally performed, tissue-based test, validated according to local regulation, from a Clinical Laboratory Improvement Amendments (CLIA)-certified US laboratory or an accredited local laboratory outside of the US. The positive METΔex14 mutation result as determined per local test must have been documented in the participant's source documents and in the CRF prior to entering main screening.
* Mandatory provision of a formalin-fixed, paraffin embedded tumor tissue sample (archival tumor block or slides, or a newly obtained tumor sample) with quality and quantity sufficient to allow assessment of METΔex14 mutation status (as defined in the study [laboratory manual]). This pertained to all participants, including those who had a METΔex14 mutation result from a local test. Tumor samples must have contained at least 10% tumor content.

  6. Participants must have progressed on one or two prior lines of systemic therapy for advanced/metastatic disease (stage IIIB/IIIC [not candidates for surgery, radiation or multi modality therapy] or IV NSCLC) and must have been docetaxel naïve and candidates for single agent chemotherapy (docetaxel). Treatment failure was defined as documented disease progression or intolerance to treatment, however, participants must have progressed on or after the last therapy before study entry.
* At least one measurable lesion as defined by RECIST 1.1
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Life expectancy of at least 3 months.

Key Exclusion Criteria:

* Prior treatment with any MET inhibitor or HGF-targeting therapy.
* Participants with symptomatic central nervous system (CNS) metastases who were neurologically unstable or had required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* Participants with known druggable molecular alterations (such as ROS1 and RET rearrangement, BRAF mutation, KRAS mutation, NTRK fusion, etc.) which might have been a candidate for alternative targeted therapies.
* Presence or history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
* Substance abuse, active infection or other severe, acute, or chronic medical or psychotic conditions or laboratory abnormalities that in the opinion of the investigator may have increased the risk associated with study participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- Novartis Investigative Site, Leuven, Belgium
- Brazil (2):
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- France (3):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
- Germany (5):
  - Novartis Investigative Site, Gauting, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Oldenburg
- Hungary (2):
  - Novartis Investigative Site, Törökbálint, Pest County
  - Novartis Investigative Site, Budapest
- India (3):
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Vellore, Tamil Nadu
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Vilnius, Lithuania
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Pulau Pinang
- Novartis Investigative Site, Nijmegen, Netherlands
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
- Russia (4):
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Pushkin Saint Petersburg
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Port Elizabeth, Western Cape, South Africa
- Novartis Investigative Site, Seoul, South Korea
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All inclusion and exclusion criteria were checked at screening.
Groups:
- Capmatinib Extension Crossover Treatment: 400 mg, capmatinib tablets, administered orally twice daily to participants treated with docetaxel who crossed over to capmatinib treatment.
Period: Randomized Treatment Phase
Arm/Group | Capmatinib | Capmatinib Extension Crossover Treatment
Started | 15 | 7
Treated | 15 | 6
Completed | 0 | 0
Not Completed | 15 | 7
Not completed — Progressive disease | 9 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Study terminated by sponsor | 3 | 0
Not completed — Death | 0 | 1
Not completed — Not treated (participant decision) | 0 | 1
Period: Extension Treatment Phase
Arm/Group | Capmatinib | Capmatinib Extension Crossover Treatment
Started | 0 | 5
Completed | 0 | 0
Not Completed | 0 | 5
Not completed — Progressive disease | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capmatinib | Docetaxel | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.26) | 65.1 (4.98) | 66.8 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 11 | 6 | 17
  Asian | 3 | 0 | 3
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Blinded Independent Review Committee (BIRC) Using RECIST v1.1
Description: Progression-free survival was defined as the time from the date of randomization to the date of the first documented progressive disease (PD) as assessed by BIRC according to RECIST 1.1, or death due to any cause. PD=At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2. PFS was censored at the date of the last adequate tumor assessment, if no PFS event was observed prior to the analysis cut-off date.
Time Frame: From randomization to the date of first documented progression or death from any cause, whichever came first, assessed up to approximately 21 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned by randomization, regardless of whether or not the treatment was administered.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
months | 6.1 [1.61 to 13.77] | 4.1 [1.22 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

2. Secondary Outcome: Overall Response (ORR) Per RECIST 1.1 by BIRC
Description: Percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR), assessed by BIRC according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
percentage of participants | 53.3 [26.59 to 78.73] | 0 [0 to 40.96]

3. Secondary Outcome: Overall Response Rate (ORR) Per RECIST 1.1 by Investigator
Description: Percentage of participants with confirmed BOR of CR or PR, assessed by local review according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
percentage of participants | 46.7 [21.27 to 73.41] | 14.3 [0.36 to 57.87]

4. Secondary Outcome: Time to Response (TTR) Per RECIST 1.1 by BIRC
Description: Time from date of randomization to first documented response of either CR or PR, which must be subsequently confirmed, assessed by BIRC according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of randomization to first documented response of either CR or PR, assessed up to approximately 21 months
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned by randomization, regardless of whether or not the treatment was administered. Data are reported for responders only.
Measure: Median (Full Range); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 8 | 0
months | 3.2 [1.2 to 15.3] |

5. Secondary Outcome: Time to Response (TTR) Per RECIST 1.1 by Investigator
Description: Time from date of randomization to first documented response of either CR or PR, which must be subsequently confirmed, assessed by local review according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of randomization to first documented response of either CR or PR, assessed up to approximately 21 months
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 7 | 1
months | 1.3 [1.2 to 15.5] | 2.8 [2.8 to 2.8]

6. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by BIRC
Description: Duration of response was defined as the time from the date of first documented response (CR or PR) to the first documented progression by BIRC per RECIST 1.1 or death due to any cause. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From first documented response to first documented progression or death due to any cause, whichever came first, assessed up to approximately 21 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 8 | 0
months | 12.6 [2.92 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with response. |

7. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 by Investigator
Description: Duration of response was defined as the time from the date of first documented response (CR or PR) to the first documented progression by local review per RECIST 1.1 or death due to any cause. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 7 | 1
months | 9.9 [2.92 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with response. | 3.1 [NA to NA] — 95% confidence interval was not calculable for a single participant.

8. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 by BIRC
Description: Disease control rate was defined as the percentage of participants with a best overall response (BOR) of confirmed CR, PR and stable disease (SD) assessed by BIRC according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD=Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
percentage of participants | 73.3 [44.90 to 92.21] | 57.1 [18.41 to 90.10]

9. Secondary Outcome: Disease Control Rate (DCR) Per RECIST 1.1 by Investigator
Description: Disease control rate was defined as the percentage of participants with a best overall response (BOR) of confirmed CR, PR and stable disease (SD) assessed by local review according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD=Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
percentage of participants | 86.7 [59.54 to 98.34] | 42.9 [9.90 to 81.59]

10. Secondary Outcome: Progression-free Survival (PFS) Per Investigator Using RECIST v1.1
Description: Progression-free survival was defined as the time from the date of randomization to the date of the first documented progressive disease (PD) as assessed by local review according to RECIST 1.1, or death due to any cause. PD=At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
months | 6.1 [2.66 to 11.10] | 3.6 [1.22 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: From randomization to death due to any cause, assessed up to approximately 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
months | 12.5 [4.30 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 13.6 [2.60 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

12. Secondary Outcome: Overall Intracranial Response Rate (OIRR)
Description: Percentage of participants with confirmed best overall intracranial response (BOIR) of CR or partial response (PR), as assessed by BIRC review per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria. Criteria for CR: Disappearance of all central nervous system (CNS) target and non-target lesions sustained for at least 4 weeks, with no new lesions, and no use of corticosteroids. PR: ≥30% decrease in the sublaterodorsal tegmental nucleus (SLD) of CNS target lesions or no new lesions or and stable to decreased corticosteroid dose.
Time Frame: Up to approximately 21 months
Population: The full analysis set - brain metastases (FAS-BM) comprised all participants in the FAS who had measurable and/or non-measurable brain metastases at baseline as determined by the BIRC and at least one post-baseline assessment. The FAS-BM was used in the analyses of intracranial anti-tumor activity per RANO-BM criteria. Data are reported for responders only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 1 | 0
Percentage of participants | 0 [0.00 to 97.50] |

13. Secondary Outcome: Duration of Intracranial Response (DOIR)
Description: Time from date of first documented intracranial response (CR or PR) to first documented intracranial progression per RANO-BM assessed by BIRC or date of death due to underlying cause of cancer.
Time Frame: From date of first documented intracranial response (CR or PR) to first documented intracranial progression, assessed up to approximately 21 months
Population: The duration of intracranial response could not be analyzed as there were no participants with intracranial response. The analysis population was all participants with intracranial response.
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Time to Intracranial Response (TTIR)
Description: Time from date of randomization to first documented intracranial response of either CR or PR, per RANO-BM criteria and assessed by BIRC, which must be subsequently confirmed.
Time Frame: From date of randomization to first documented intracranial response of either CR or PR, assessed up to approximately 21 months
Population: The median time to intracranial response was not evaluable in both treatment arms as there were no responders.
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Intracranial Disease Control Rate (IDCR)
Description: Percentage of participants with a BOR of confirmed CR, PR and stable disease (SD) (or non-CR/non-PD) per RANO-BM, assessed by BIRC. Criteria for CR: Disappearance of all central nervous system (CNS) target and non-target lesions sustained for at least 4 weeks, with no new lesions, and no use of corticosteroids. PR: ≥30% decrease in the sublaterodorsal tegmental nucleus (SLD) of CNS target lesions or no new lesions or and stable to decreased corticosteroid dose.
Time Frame: Up to approximately 21 months
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 1 | 0
percentage of participants | 100 [2.50 to 100] |

16. Secondary Outcome: Plasma Capmatinib Concentration
Description: Plasma concentrations of capmatinib. Blood samples were collected at indicated time points for pharmacokinetic analysis.
Time Frame: Cycle (C) 1 Day (D) 15 pre-dose, 1 and 4 hours post-dose, C3 D1 pre-dose. Each cycle duration was 21 days.
Population: The pharmacokinetic analysis set (PAS) included all participants who received at least one dose of capmatinib and had at least one steady state evaluable post-baseline capmatinib concentration measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Capmatinib
Number analyzed (Participants) | 14
μg/mL
  Cycle 1, Day 15, 0 hour n=12: number analyzed (Participants) | 12
  Cycle 1, Day 15, 0 hour n=12 | 496 (97.3)
  Cycle 1, Day 15, 1 hour n=10: number analyzed (Participants) | 10
  Cycle 1, Day 15, 1 hour n=10 | 1330 (214.6)
  Cycle 1, Day 15, 4 hours n=11: number analyzed (Participants) | 11
  Cycle 1, Day 15, 4 hours n=11 | 2680 (131.1)
  Cycle 3, Day 1, 0 hour n=10: number analyzed (Participants) | 10
  Cycle 3, Day 1, 0 hour n=10 | 243 (140.6)

17. Secondary Outcome: Change From Baseline in Score as Per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. The questionnaire is composed of both multi-item scales and single-item measures based on the participants experience over the past week. These include five domains (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact) and a global health status/HRQoL scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. CFB = change from baseline.
Time Frame: Baseline, Cycle (C) 3, Day (D) 1 and then every 6 weeks up to approximately 21 months, end of treatment. Each cycle duration was 21 days.
Population: The full analysis set (FAS) comprised all participants to whom study treatment was assigned by randomization, regardless of whether or not the treatment was administered. Data are reported for participants with baseline and respective post-baseline measurements.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
score on a scale
  Global Health Status CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Global Health Status CFB at Cycle 3, Day 1 n=12,4 | 17.4 (18.96) | 4.2 (14.43)
  Global Health Status CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Global Health Status CFB at Cycle 5, Day 1 n=8,3 | 14.6 (22.16) | 8.3 (14.43)
  Global Health Status CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Global Health Status CFB at Cycle 7, Day 1 n=8,1 | 15.6 (16.33) | -8.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Global Health Status CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Global Health Status CFB at Cycle 9, Day 1 n=7,2 | 9.5 (16.96) | 0.0 (11.79)
  Global Health Status CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Global Health Status CFB at Cycle 11, Day 1 n=7,0 | 3.6 (15.85) |
  Global Health Status CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Global Health Status CFB at Cycle 13, Day 1 n=5,0 | 25.0 (10.21) |
  Global Health Status CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Global Health Status CFB at Cycle 15, Day 1 n=5,0 | 10.0 (10.87) |
  Global Health Status CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Global Health Status CFB at Cycle 17, Day 1 n=4,0 | 18.8 (10.49) |
  Global Health Status CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Global Health Status CFB at Cycle 19, Day 1 n=5,0 | -1.7 (19.00) |
  Global Health Status CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Global Health Status CFB at Cycle 21, Day 1 n=4,0 | 0.0 (0.00) |
  Global Health Status CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Global Health Status CFB at Cycle 23, Day 1 n=2,0 | -8.3 (11.79) |
  Global Health Status CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Global Health Status CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Global Health Status CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Global Health Status CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Global Health Status CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Global Health Status CFB at Cycle 29, Day 1 n=2,0 | -29.2 (29.46) |
  Physical Functioning CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Physical Functioning CFB at Cycle 3, Day 1 n=12,4 | 11.1 (24.01) | -1.7 (6.38)
  Physical Functioning CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Physical Functioning CFB at Cycle 5, Day 1 n=8,3 | 15.0 (21.89) | -13.3 (23.09)
  Physical Functioning CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Physical Functioning CFB at Cycle 7, Day 1 n=8,1 | 4.2 (26.41) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Physical Functioning CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Physical Functioning CFB at Cycle 9, Day 1 n=7,2 | 7.6 (22.25) | 3.3 (14.14)
  Physical Functioning CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Physical Functioning CFB at Cycle 11, Day 1 n=7,0 | -1.9 (25.74) |
  Physical Functioning CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Physical Functioning CFB at Cycle 13, Day 1 n=5,0 | 5.3 (25.99) |
  Physical Functioning CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Physical Functioning CFB at Cycle 15, Day 1 n=5,0 | -1.3 (15.92) |
  Physical Functioning CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Physical Functioning CFB at Cycle 17, Day 1 n=4,0 | -5.0 (13.74) |
  Physical Functioning CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Physical Functioning CFB at Cycle 19, Day 1 n=5,0 | -2.7 (32.52) |
  Physical Functioning CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Physical Functioning CFB at Cycle 21, Day 1 n=4,0 | 5.0 (10.00) |
  Physical Functioning CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Physical Functioning CFB at Cycle 23, Day 1 n=2,0 | 0.0 (9.43) |
  Physical Functioning CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Physical Functioning CFB at Cycle 25, Day 1 n=2,0 | 13.3 (9.43) |
  Physical Functioning CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Physical Functioning CFB at Cycle 27, Day 1 n=2,0 | 3.3 (4.71) |
  Physical Functioning CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Physical Functioning CFB at Cycle 29, Day 1 n=2,0 | 0.0 (28.28) |
  Role Functioning CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Role Functioning CFB at Cycle 3, Day 1 n=12,4 | 20.8 (22.61) | -4.2 (20.97)
  Role Functioning CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Role Functioning CFB at Cycle 5, Day 1 n=8,3 | 20.8 (29.21) | -5.6 (25.46)
  Role Functioning CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Role Functioning CFB at Cycle 7, Day 1 n=8,1 | 18.8 (28.78) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Role Functioning CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Role Functioning CFB at Cycle 9, Day 1 n=7,2 | 14.3 (22.42) | -8.3 (11.79)
  Role Functioning CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Role Functioning CFB at Cycle 11, Day 1 n=7,0 | 7.1 (26.97) |
  Role Functioning CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Role Functioning CFB at Cycle 13, Day 1 n=5,0 | 13.3 (21.73) |
  Role Functioning CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Role Functioning CFB at Cycle 15, Day 1 n=5,0 | 26.7 (19.00) |
  Role Functioning CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Role Functioning CFB at Cycle 17, Day 1 n=4,0 | 0.0 (13.61) |
  Role Functioning CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Role Functioning CFB at Cycle 19, Day 1 n=5,0 | 16.7 (50.00) |
  Role Functioning CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Role Functioning CFB at Cycle 21, Day 1 n=4,0 | 8.3 (16.67) |
  Role Functioning CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Role Functioning CFB at Cycle 23, Day 1 n=2,0 | 8.3 (11.79) |
  Role Functioning CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Role Functioning CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Role Functioning CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Role Functioning CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Role Functioning CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Role Functioning CFB at Cycle 29, Day 1 n=2,0 | 0.0 (47.14) |
  Emotional Functioning CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Emotional Functioning CFB at Cycle 3, Day 1 n=12,4 | 15.3 (32.14) | 2.1 (7.98)
  Emotional Functioning CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Emotional Functioning CFB at Cycle 5, Day 1 n=8,3 | 15.6 (31.32) | 11.1 (17.35)
  Emotional Functioning CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Emotional Functioning CFB at Cycle 7, Day 1 n=8,1 | 12.5 (34.21) | -16.7 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Emotional Functioning CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Emotional Functioning CFB at Cycle 9, Day 1 n=7,2 | 8.3 (36.00) | -8.3 (11.79)
  Emotional Functioning CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Emotional Functioning CFB at Cycle 11, Day 1 n=7,0 | 1.2 (23.29) |
  Emotional Functioning CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Emotional Functioning CFB at Cycle 13, Day 1 n=5,0 | 18.3 (25.28) |
  Emotional Functioning CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Emotional Functioning CFB at Cycle 15, Day 1 n=5,0 | 16.7 (19.54) |
  Emotional Functioning CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Emotional Functioning CFB at Cycle 17, Day 1 n=4,0 | 8.3 (11.79) |
  Emotional Functioning CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Emotional Functioning CFB at Cycle 19, Day 1 n=5,0 | 15.0 (21.57) |
  Emotional Functioning CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Emotional Functioning CFB at Cycle 21, Day 1 n=4,0 | 16.7 (15.21) |
  Emotional Functioning CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Emotional Functioning CFB at Cycle 23, Day 1 n=2,0 | 0.0 (11.79) |
  Emotional Functioning CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Emotional Functioning CFB at Cycle 25, Day 1 n=2,0 | 8.3 (47.14) |
  Emotional Functioning CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Emotional Functioning CFB at Cycle 27, Day 1 n=2,0 | -8.3 (23.57) |
  Emotional Functioning CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Emotional Functioning CFB at Cycle 29, Day 1 n=2,0 | 8.3 (35.36) |
  Cognitive Functioning CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Cognitive Functioning CFB at Cycle 3, Day 1 n=12,4 | 12.5 (23.70) | -8.3 (9.62)
  Cognitive Functioning CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Cognitive Functioning CFB at Cycle 5, Day 1 n=8,3 | 6.3 (29.46) | 0.0 (16.67)
  Cognitive Functioning CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Cognitive Functioning CFB at Cycle 7, Day 1 n=8,1 | 6.3 (33.26) | 16.7 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Cognitive Functioning CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Cognitive Functioning CFB at Cycle 9, Day 1 n=7,2 | 7.1 (21.21) | 8.3 (11.79)
  Cognitive Functioning CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Cognitive Functioning CFB at Cycle 11, Day 1 n=7,0 | 4.8 (23.00) |
  Cognitive Functioning CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Cognitive Functioning CFB at Cycle 13, Day 1 n=5,0 | 20.0 (18.26) |
  Cognitive Functioning CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Cognitive Functioning CFB at Cycle 15, Day 1 n=5,0 | 16.7 (16.67) |
  Cognitive Functioning CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Cognitive Functioning CFB at Cycle 17, Day 1 n=4,0 | 8.3 (21.52) |
  Cognitive Functioning CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Cognitive Functioning CFB at Cycle 19, Day 1 n=5,0 | 16.7 (28.87) |
  Cognitive Functioning CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Cognitive Functioning CFB at Cycle 21, Day 1 n=4,0 | 0.0 (13.61) |
  Cognitive Functioning CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cognitive Functioning CFB at Cycle 23, Day 1 n=2,0 | 8.3 (35.36) |
  Cognitive Functioning CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cognitive Functioning CFB at Cycle 25, Day 1 n=2,0 | 0.0 (47.14) |
  Cognitive Functioning CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cognitive Functioning CFB at Cycle 27, Day 1 n=2,0 | -8.3 (35.36) |
  Cognitive Functioning CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Cognitive Functioning CFB at Cycle 29, Day 1 n=2,0 | 41.7 (11.79) |
  Social Functioning CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Social Functioning CFB at Cycle 3, Day 1 n=12,4 | 18.1 (37.91) | -4.2 (25.00)
  Social Functioning CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Social Functioning CFB at Cycle 5, Day 1 n=8,3 | 12.5 (44.32) | -22.2 (19.25)
  Social Functioning CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Social Functioning CFB at Cycle 7, Day 1 n=8,1 | -2.1 (37.20) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Social Functioning CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Social Functioning CFB at Cycle 9, Day 1 n=7,2 | 0.0 (33.33) | 0.0 (47.14)
  Social Functioning CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Social Functioning CFB at Cycle 11, Day 1 n=7,0 | -2.4 (35.26) |
  Social Functioning CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Social Functioning CFB at Cycle 13, Day 1 n=5,0 | 23.3 (25.28) |
  Social Functioning CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Social Functioning CFB at Cycle 15, Day 1 n=5,0 | 10.0 (25.28) |
  Social Functioning CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Social Functioning CFB at Cycle 17, Day 1 n=4,0 | 16.7 (23.57) |
  Social Functioning CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Social Functioning CFB at Cycle 19, Day 1 n=5,0 | -13.3 (13.94) |
  Social Functioning CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Social Functioning CFB at Cycle 21, Day 1 n=4,0 | -16.7 (13.61) |
  Social Functioning CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Social Functioning CFB at Cycle 23, Day 1 n=2,0 | -8.3 (11.79) |
  Social Functioning CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Social Functioning CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Social Functioning CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Social Functioning CFB at Cycle 27, Day 1 n=2,0 | -16.7 (23.57) |
  Social Functioning CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Social Functioning CFB at Cycle 29, Day 1 n=2,0 | -8.3 (11.79) |
  Fatigue CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Fatigue CFB at Cycle 3, Day 1 n=12,4 | -11.1 (31.43) | -11.1 (9.07)
  Fatigue CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Fatigue CFB at Cycle 5, Day 1 n=8,3 | -12.5 (27.50) | -14.8 (23.13)
  Fatigue CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Fatigue CFB at Cycle 7, Day 1 n=8,1 | -12.5 (29.36) | -22.2 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Fatigue CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Fatigue CFB at Cycle 9, Day 1 n=7,2 | -12.7 (25.20) | -11.1 (15.71)
  Fatigue CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Fatigue CFB at Cycle 11, Day 1 n=7,0 | -7.9 (27.75) |
  Fatigue CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Fatigue CFB at Cycle 13, Day 1 n=5,0 | -13.3 (27.67) |
  Fatigue CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Fatigue CFB at Cycle 15, Day 1 n=5,0 | -15.6 (16.85) |
  Fatigue CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Fatigue CFB at Cycle 17, Day 1 n=4,0 | -5.6 (14.34) |
  Fatigue CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Fatigue CFB at Cycle 19, Day 1 n=5,0 | -4.4 (26.76) |
  Fatigue CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Fatigue CFB at Cycle 21, Day 1 n=4,0 | -11.1 (15.71) |
  Fatigue CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Fatigue CFB at Cycle 23, Day 1 n=2,0 | 0.0 (0.0) |
  Fatigue CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Fatigue CFB at Cycle 25, Day 1 n=2,0 | -16.7 (23.57) |
  Fatigue CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Fatigue CFB at Cycle 27, Day 1 n=2,0 | 5.6 (7.86) |
  Fatigue CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Fatigue CFB at Cycle 29, Day 1 n=2,0 | 11.1 (31.43) |
  Nausea and Vomiting CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Nausea and Vomiting CFB at Cycle 3, Day 1 n=12,4 | -1.4 (21.86) | 0.0 (0.00)
  Nausea and Vomiting CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Nausea and Vomiting CFB at Cycle 5, Day 1 n=8,3 | -6.3 (26.63) | 11.1 (9.62)
  Nausea and Vomiting CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Nausea and Vomiting CFB at Cycle 7, Day 1 n=8,1 | 20.8 (39.59) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Nausea and Vomiting CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Nausea and Vomiting CFB at Cycle 9, Day 1 n=7,2 | 0.0 (23.57) | 0.0 (0.00)
  Nausea and Vomiting CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Nausea and Vomiting CFB at Cycle 11, Day 1 n=7,0 | 4.8 (28.41) |
  Nausea and Vomiting CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Nausea and Vomiting CFB at Cycle 13, Day 1 n=5,0 | -3.3 (7.45) |
  Nausea and Vomiting CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Nausea and Vomiting CFB at Cycle 15, Day 1 n=5,0 | 0.0 (16.67) |
  Nausea and Vomiting CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Nausea and Vomiting CFB at Cycle 17, Day 1 n=4,0 | 8.3 (31.91) |
  Nausea and Vomiting CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Nausea and Vomiting CFB at Cycle 19, Day 1 n=5,0 | 20.0 (49.16) |
  Nausea and Vomiting CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Nausea and Vomiting CFB at Cycle 21, Day 1 n=4,0 | 20.8 (34.36) |
  Nausea and Vomiting CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Nausea and Vomiting CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Nausea and Vomiting CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Nausea and Vomiting CFB at Cycle 25, Day 1 n=2,0 | 8.3 (35.36) |
  Nausea and Vomiting CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Nausea and Vomiting CFB at Cycle 27, Day 1 n=2,0 | 16.7 (47.14) |
  Nausea and Vomiting CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Nausea and Vomiting CFB at Cycle 29, Day 1 n=2,0 | 8.3 (35.36) |
  Pain CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Pain CFB at Cycle 3, Day 1 n=12,4 | -4.2 (41.51) | -25.0 (16.67)
  Pain CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Pain CFB at Cycle 5, Day 1 n=8,3 | -2.1 (31.42) | 5.6 (38.49)
  Pain CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Pain CFB at Cycle 7, Day 1 n=8,1 | -4.2 (42.49) | -16.7 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Pain CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Pain CFB at Cycle 9, Day 1 n=7,2 | -4.8 (29.99) | 0.0 (0.00)
  Pain CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Pain CFB at Cycle 11, Day 1 n=7,0 | 4.8 (50.66) |
  Pain CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain CFB at Cycle 13, Day 1 n=5,0 | 0.0 (54.01) |
  Pain CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain CFB at Cycle 15, Day 1 n=5,0 | -6.7 (40.14) |
  Pain CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain CFB at Cycle 17, Day 1 n=4,0 | 12.5 (77.43) |
  Pain CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain CFB at Cycle 19, Day 1 n=5,0 | 6.7 (63.03) |
  Pain CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain CFB at Cycle 21, Day 1 n=4,0 | 4.2 (43.83) |
  Pain CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain CFB at Cycle 23, Day 1 n=2,0 | 25.0 (35.36) |
  Pain CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain CFB at Cycle 25, Day 1 n=2,0 | 16.7 (70.71) |
  Pain CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain CFB at Cycle 27, Day 1 n=2,0 | 33.3 (47.14) |
  Pain CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain CFB at Cycle 29, Day 1 n=2,0 | -16.7 (23.57) |
  Dyspnea CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Dyspnea CFB at Cycle 3, Day 1 n=12,4 | -13.9 (33.21) | 0.0 (0.00)
  Dyspnea CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Dyspnea CFB at Cycle 5, Day 1 n=8,3 | -12.5 (30.54) | 11.1 (19.25)
  Dyspnea CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Dyspnea CFB at Cycle 7, Day 1 n=8,1 | -4.2 (27.82) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Dyspnea CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Dyspnea CFB at Cycle 9, Day 1 n=7,2 | -4.8 (23.00) | 16.7 (23.57)
  Dyspnea CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Dyspnea CFB at Cycle 11, Day 1 n=7,0 | 14.3 (37.80) |
  Dyspnea CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dyspnea CFB at Cycle 13, Day 1 n=5,0 | 6.7 (27.89) |
  Dyspnea CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dyspnea CFB at Cycle 15, Day 1 n=5,0 | 20.0 (29.81) |
  Dyspnea CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Dyspnea CFB at Cycle 17, Day 1 n=4,0 | 8.3 (16.67) |
  Dyspnea CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dyspnea CFB at Cycle 19, Day 1 n=5,0 | 13.3 (29.81) |
  Dyspnea CFB at Cycle 21, Day 1 n=: number analyzed (Participants) | 4 | 0
  Dyspnea CFB at Cycle 21, Day 1 n= | 16.7 (43.03) |
  Dyspnea CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Dyspnea CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Dyspnea CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Dyspnea CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Insomnia CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Insomnia CFB at Cycle 3, Day 1 n=12,4 | -13.9 (26.43) | 8.3 (31.91)
  Insomnia CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Insomnia CFB at Cycle 5, Day 1 n=8,3 | 0.0 (25.20) | -22.2 (19.25)
  Insomnia CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Insomnia CFB at Cycle 7, Day 1 n=8,1 | -8.3 (34.50) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Insomnia CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Insomnia CFB at Cycle 9, Day 1 n=7,2 | -4.8 (35.63) | 0.0 (0.00)
  Insomnia CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Insomnia CFB at Cycle 11, Day 1 n=7,0 | 0.0 (38.49) |
  Insomnia CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Insomnia CFB at Cycle 13, Day 1 n=5,0 | 0.0 (33.33) |
  Insomnia CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Insomnia CFB at Cycle 15, Day 1 n=5,0 | -13.3 (38.01) |
  Insomnia CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Insomnia CFB at Cycle 17, Day 1 n=4,0 | 16.7 (43.03) |
  Insomnia CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Insomnia CFB at Cycle 19, Day 1 n=5,0 | -6.7 (49.44) |
  Insomnia CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Insomnia CFB at Cycle 21, Day 1 n=4,0 | 0.0 (72.01) |
  Insomnia CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Insomnia CFB at Cycle 23, Day 1 n=2,0 | 0.0 (0.00) |
  Insomnia CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Insomnia CFB at Cycle 25, Day 1 n=2,0 | -16.7 (23.57) |
  Insomnia CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Insomnia CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Insomnia CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Insomnia CFB at Cycle 29, Day 1 n=2,0 | 16.7 (70.71) |
  Appetite Loss CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Appetite Loss CFB at Cycle 3, Day 1 n=12,4 | -16.7 (38.92) | -8.3 (16.67)
  Appetite Loss CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Appetite Loss CFB at Cycle 5, Day 1 n=8,3 | 4.2 (41.55) | -11.1 (19.25)
  Appetite Loss CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Appetite Loss CFB at Cycle 7, Day 1 n=8,1 | -12.5 (24.80) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Appetite Loss CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Appetite Loss CFB at Cycle 9, Day 1 n=7,2 | -19.0 (32.53) | 0.0 (47.14)
  Appetite Loss CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Appetite Loss CFB at Cycle 11, Day 1 n=7,0 | -14.3 (42.41) |
  Appetite Loss CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Appetite Loss CFB at Cycle 13, Day 1 n=5,0 | -40.0 (36.51) |
  Appetite Loss CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Appetite Loss CFB at Cycle 15, Day 1 n=5,0 | -33.3 (47.14) |
  Appetite Loss CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Appetite Loss CFB at Cycle 17, Day 1 n=4,0 | -33.3 (47.14) |
  Appetite Loss CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Appetite Loss CFB at Cycle 19, Day 1 n=5,0 | -13.3 (73.03) |
  Appetite Loss CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Appetite Loss CFB at Cycle 21, Day 1 n=4,0 | -33.3 (47.14) |
  Appetite Loss CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Appetite Loss CFB at Cycle 23, Day 1 n=2,0 | -16.7 (23.57) |
  Appetite Loss CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Appetite Loss CFB at Cycle 25, Day 1 n=2,0 | -16.7 (23.57) |
  Appetite Loss CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Appetite Loss CFB at Cycle 27, Day 1 n=2,0 | -33.3 (0.00) |
  Appetite Loss CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Appetite Loss CFB at Cycle 29, Day 1 n=2,0 | -33.3 (0.00) |
  Constipation CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Constipation CFB at Cycle 3, Day 1 n=12,4 | 2.8 (38.82) | -16.7 (19.25)
  Constipation CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Constipation CFB at Cycle 5, Day 1 n=8,3 | -12.5 (35.36) | 0.0 (33.33)
  Constipation CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Constipation CFB at Cycle 7, Day 1 n=8,1 | -4.2 (54.74) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Constipation CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Constipation CFB at Cycle 9, Day 1 n=7,2 | 14.3 (26.23) | -33.3 (0.00)
  Constipation CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Constipation CFB at Cycle 11, Day 1 n=7,0 | -4.8 (44.84) |
  Constipation CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Constipation CFB at Cycle 13, Day 1 n=5,0 | -20.0 (44.72) |
  Constipation CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Constipation CFB at Cycle 15, Day 1 n=5,0 | -6.7 (54.77) |
  Constipation CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Constipation CFB at Cycle 17, Day 1 n=4,0 | -16.7 (57.74) |
  Constipation CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Constipation CFB at Cycle 19, Day 1 n=5,0 | -26.7 (43.46) |
  Constipation CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Constipation CFB at Cycle 21, Day 1 n=4,0 | -16.7 (57.74) |
  Constipation CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Constipation CFB at Cycle 23, Day 1 n=2,0 | 33.3 (0.00) |
  Constipation CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Constipation CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Constipation CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Constipation CFB at Cycle 27, Day 1 n=2,0 | 16.7 (23.57) |
  Constipation CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Constipation CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Diarrhea CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Diarrhea CFB at Cycle 3, Day 1 n=12,4 | 0.0 (24.62) | 0.0 (0.00)
  Diarrhea CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Diarrhea CFB at Cycle 5, Day 1 n=8,3 | -4.2 (11.79) | -22.2 (38.49)
  Diarrhea CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Diarrhea CFB at Cycle 7, Day 1 n=8,1 | 0.0 (17.82) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Diarrhea CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Diarrhea CFB at Cycle 9, Day 1 n=7,2 | 14.3 (17.82) | 0.0 (0.00)
  Diarrhea CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Diarrhea CFB at Cycle 11, Day 1 n=7,0 | 4.8 (12.60) |
  Diarrhea CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Diarrhea CFB at Cycle 13, Day 1 n=5,0 | 0.0 (0.00) |
  Diarrhea CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Diarrhea CFB at Cycle 15, Day 1 n=5,0 | 6.7 (14.91) |
  Diarrhea CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Diarrhea CFB at Cycle 17, Day 1 n=4,0 | 16.7 (33.33) |
  Diarrhea CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Diarrhea CFB at Cycle 19, Day 1 n=5,0 | 13.3 (29.81) |
  Diarrhea CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Diarrhea CFB at Cycle 21, Day 1 n=4,0 | 8.3 (16.67) |
  Diarrhea CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Diarrhea CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Diarrhea CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Diarrhea CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Diarrhea CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Diarrhea CFB at Cycle 27, Day 1 n=2,0 | 16.7 (23.57) |
  Diarrhea CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Diarrhea CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Financial Difficulties CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Financial Difficulties CFB at Cycle 3, Day 1 n=12,4 | -2.8 (26.43) | 0.0 (0.00)
  Financial Difficulties CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Financial Difficulties CFB at Cycle 5, Day 1 n=8,3 | -8.3 (29.55) | -11.1 (19.25)
  Financial Difficulties CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Financial Difficulties CFB at Cycle 7, Day 1 n=8,1 | -4.2 (21.36) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Financial Difficulties CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Financial Difficulties CFB at Cycle 9, Day 1 n=7,2 | 0.0 (33.33) | -33.3 (47.14)
  Financial Difficulties CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Financial Difficulties CFB at Cycle 11, Day 1 n=7,0 | 0.0 (19.25) |
  Financial Difficulties CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Financial Difficulties CFB at Cycle 13, Day 1 n=5,0 | 0.0 (23.57) |
  Financial Difficulties CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Financial Difficulties CFB at Cycle 15, Day 1 n=5,0 | 13.3 (18.26) |
  Financial Difficulties CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Financial Difficulties CFB at Cycle 17, Day 1 n=4,0 | -8.3 (31.91) |
  Financial Difficulties CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Financial Difficulties CFB at Cycle 19, Day 1 n=5,0 | 13.3 (29.81) |
  Financial Difficulties CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Financial Difficulties CFB at Cycle 21, Day 1 n=4,0 | 25.0 (16.67) |
  Financial Difficulties CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Financial Difficulties CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Financial Difficulties CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Financial Difficulties CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Financial Difficulties CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Financial Difficulties CFB at Cycle 27, Day 1 n=2,0 | 33.3 (0.00) |
  Financial Difficulties CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Financial Difficulties CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |

18. Secondary Outcome: Change From Baseline in Score as Per European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Lung Cancer Module (QLQ-LC13)
Description: EORTC QLQ-LC13 is a 13-item lung cancer specific questionnaire. The assessments here included coughing, hemoptysis, dyspnea, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, and pain in other parts and were based on their presence over the previous week. All but the pain domain were scored on a 4 point Likert scale ranging from "not at all" to "very much." Pain was scored based on its presence, yes or no. Scores were averaged and transformed to 0 to 100. A higher score indicated a higher presence of symptoms. CFB = change from baseline.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
score on a scale
  Coughing CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Coughing CFB at Cycle 3, Day 1 n=12,4 | -19.4 (26.43) | 16.7 (19.25)
  Coughing CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Coughing CFB at Cycle 5, Day 1 n=8,3 | -8.3 (23.57) | 11.1 (19.25)
  Coughing CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Coughing CFB at Cycle 7, Day 1 n=8,1 | -20.8 (24.80) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Coughing CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Coughing CFB at Cycle 9, Day 1 n=7,2 | -23.8 (25.20) | 0.0 (0.00)
  Coughing CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Coughing CFB at Cycle 11, Day 1 n=7,0 | -9.5 (37.09) |
  Coughing CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Coughing CFB at Cycle 13, Day 1 n=5,0 | -20.0 (29.81) |
  Coughing CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Coughing CFB at Cycle 15, Day 1 n=5,0 | -6.7 (36.51) |
  Coughing CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Coughing CFB at Cycle 17, Day 1 n=4,0 | 0.0 (0.00) |
  Coughing CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Coughing CFB at Cycle 19, Day 1 n=5,0 | -6.7 (14.91) |
  Coughing CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Coughing CFB at Cycle 21, Day 1 n=4,0 | -8.3 (41.94) |
  Coughing CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Coughing CFB at Cycle 23, Day 1 n=2,0 | 0.0 (0.00) |
  Coughing CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Coughing CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Coughing CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Coughing CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Coughing CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Coughing CFB at Cycle 29, Day 1 n=2,0 | -16.7 (23.57) |
  Hemoptysis CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Hemoptysis CFB at Cycle 3, Day 1 n=12,4 | 0.0 (0.00) | 8.3 (16.67)
  Hemoptysis CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Hemoptysis CFB at Cycle 5, Day 1 n=8,3 | 0.0 (0.00) | 0.0 (0.00)
  Hemoptysis CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Hemoptysis CFB at Cycle 7, Day 1 n=8,1 | 4.2 (11.79) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Hemoptysis CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Hemoptysis CFB at Cycle 9, Day 1 n=7,2 | 0.0 (0.00) | 0.0 (0.00)
  Hemoptysis CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Hemoptysis CFB at Cycle 11, Day 1 n=7,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Hemoptysis CFB at Cycle 13, Day 1 n=5,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Hemoptysis CFB at Cycle 15, Day 1 n=5,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Hemoptysis CFB at Cycle 17, Day 1 n=4,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Hemoptysis CFB at Cycle 19, Day 1 n=5,0 | 13.3 (29.81) |
  Hemoptysis CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Hemoptysis CFB at Cycle 21, Day 1 n=4,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Hemoptysis CFB at Cycle 23, Day 1 n=2,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Hemoptysis CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Hemoptysis CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Hemoptysis CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Hemoptysis CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Dyspnea CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Dyspnea CFB at Cycle 3, Day 1 n=12,4 | -20.4 (21.10) | 0.0 (9.07)
  Dyspnea CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Dyspnea CFB at Cycle 5, Day 1 n=8,3 | -18.1 (17.76) | 14.8 (16.97)
  Dyspnea CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Dyspnea CFB at Cycle 7, Day 1 n=8,1 | -8.3 (29.55) | 11.1 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Dyspnea CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Dyspnea CFB at Cycle 9, Day 1 n=7,2 | -14.3 (33.16) | 16.7 (23.57)
  Dyspnea CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Dyspnea CFB at Cycle 11, Day 1 n=7,0 | -4.8 (32.62) |
  Dyspnea CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dyspnea CFB at Cycle 13, Day 1 n=5,0 | -13.3 (31.82) |
  Dyspnea CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dyspnea CFB at Cycle 15, Day 1 n=5,0 | -11.1 (27.22) |
  Dyspnea CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Dyspnea CFB at Cycle 17, Day 1 n=4,0 | 0.0 (9.07) |
  Dyspnea CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dyspnea CFB at Cycle 19, Day 1 n=5,0 | 6.7 (30.02) |
  Dyspnea CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Dyspnea CFB at Cycle 21, Day 1 n=4,0 | -2.8 (36.71) |
  Dyspnea CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 23, Day 1 n=2,0 | -5.6 (7.86) |
  Dyspnea CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 25, Day 1 n=2,0 | -5.6 (7.86) |
  Dyspnea CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 27, Day 1 n=2,0 | -5.6 (7.86) |
  Dyspnea CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dyspnea CFB at Cycle 29, Day 1 n=2,0 | 0.0 (15.71) |
  Sore Mouth CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Sore Mouth CFB at Cycle 3, Day 1 n=12,4 | -8.3 (25.13) | 0.0 (0.00)
  Sore Mouth CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Sore Mouth CFB at Cycle 5, Day 1 n=8,3 | -4.2 (11.79) | 0.0 (0.00)
  Sore Mouth CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Sore Mouth CFB at Cycle 7, Day 1 n=8,1 | -4.2 (27.82) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Sore Mouth CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Sore Mouth CFB at Cycle 9, Day 1 n=7,2 | 9.5 (16.27) | 16.7 (23.57)
  Sore Mouth CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Sore Mouth CFB at Cycle 11, Day 1 n=7,0 | 9.5 (16.27) |
  Sore Mouth CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Sore Mouth CFB at Cycle 13, Day 1 n=5,0 | 13.3 (18.26) |
  Sore Mouth CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Sore Mouth CFB at Cycle 15, Day 1 n=5,0 | 13.3 (29.81) |
  Sore Mouth CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Sore Mouth CFB at Cycle 17, Day 1 n=4,0 | 16.7 (33.33) |
  Sore Mouth CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Sore Mouth CFB at Cycle 19, Day 1 n=5,0 | 33.3 (33.33) |
  Sore Mouth CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Sore Mouth CFB at Cycle 21, Day 1 n=4,0 | 8.3 (16.67) |
  Sore Mouth CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Sore Mouth CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Sore Mouth CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Sore Mouth CFB at Cycle 25, Day 1 n=2,0 | 33.3 (47.14) |
  Sore Mouth CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Sore Mouth CFB at Cycle 27, Day 1 n=2,0 | 33.3 (47.14) |
  Sore Mouth CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Sore Mouth CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Dysphagia CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Dysphagia CFB at Cycle 3, Day 1 n=12,4 | 0.0 (14.21) | 0.0 (0.00)
  Dysphagia CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Dysphagia CFB at Cycle 5, Day 1 n=8,3 | 8.3 (23.57) | 0.0 (0.00)
  Dysphagia CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Dysphagia CFB at Cycle 7, Day 1 n=8,1 | 12.5 (24.80) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Dysphagia CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Dysphagia CFB at Cycle 9, Day 1 n=7,2 | 4.8 (12.60) | 0.0 (0.00)
  Dysphagia CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Dysphagia CFB at Cycle 11, Day 1 n=7,0 | 9.5 (16.27) |
  Dysphagia CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dysphagia CFB at Cycle 13, Day 1 n=5,0 | 6.7 (14.91) |
  Dysphagia CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dysphagia CFB at Cycle 15, Day 1 n=5,0 | 13.3 (18.26) |
  Dysphagia CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Dysphagia CFB at Cycle 17, Day 1 n=4,0 | 25.0 (31.91) |
  Dysphagia CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Dysphagia CFB at Cycle 19, Day 1 n=5,0 | 20.0 (18.26) |
  Dysphagia CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Dysphagia CFB at Cycle 21, Day 1 n=4,0 | 25.0 (31.91) |
  Dysphagia CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dysphagia CFB at Cycle 23, Day 1 n=2,0 | 33.3 (47.14) |
  Dysphagia CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dysphagia CFB at Cycle 25, Day 1 n=2,0 | 33.3 (47.14) |
  Dysphagia CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dysphagia CFB at Cycle 27, Day 1 n=2,0 | 33.3 (47.14) |
  Dysphagia CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Dysphagia CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Peripheral Neuropathy CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Peripheral Neuropathy CFB at Cycle 3, Day 1 n=12,4 | 13.9 (26.43) | 8.3 (31.91)
  Peripheral Neuropathy CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Peripheral Neuropathy CFB at Cycle 5, Day 1 n=8,3 | -4.2 (11.79) | 11.1 (38.49)
  Peripheral Neuropathy CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Peripheral Neuropathy CFB at Cycle 7, Day 1 n=8,1 | 20.8 (17.25) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Peripheral Neuropathy CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Peripheral Neuropathy CFB at Cycle 9, Day 1 n=7,2 | 28.6 (23.00) | -16.7 (23.57)
  Peripheral Neuropathy CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Peripheral Neuropathy CFB at Cycle 11, Day 1 n=7,0 | 14.3 (17.82) |
  Peripheral Neuropathy CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Peripheral Neuropathy CFB at Cycle 13, Day 1 n=5,0 | 13.3 (18.26) |
  Peripheral Neuropathy CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Peripheral Neuropathy CFB at Cycle 15, Day 1 n=5,0 | 6.7 (14.91) |
  Peripheral Neuropathy CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Peripheral Neuropathy CFB at Cycle 17, Day 1 n=4,0 | 8.3 (16.67) |
  Peripheral Neuropathy CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Peripheral Neuropathy CFB at Cycle 19, Day 1 n=5,0 | 26.7 (43.46) |
  Peripheral Neuropathy CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Peripheral Neuropathy CFB at Cycle 21, Day 1 n=4,0 | 25.0 (31.91) |
  Peripheral Neuropathy CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Peripheral Neuropathy CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Peripheral Neuropathy CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Peripheral Neuropathy CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Peripheral Neuropathy CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Peripheral Neuropathy CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Peripheral Neuropathy CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Peripheral Neuropathy CFB at Cycle 29, Day 1 n=2,0 | 16.7 (23.57) |
  Alopecia CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Alopecia CFB at Cycle 3, Day 1 n=12,4 | -8.3 (20.72) | 41.7 (41.94)
  Alopecia CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Alopecia CFB at Cycle 5, Day 1 n=8,3 | -16.7 (17.82) | 22.2 (19.25)
  Alopecia CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Alopecia CFB at Cycle 7, Day 1 n=8,1 | 0.0 (25.20) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Alopecia CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Alopecia CFB at Cycle 9, Day 1 n=7,2 | 0.0 (19.25) | 0.0 (47.14)
  Alopecia CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Alopecia CFB at Cycle 11, Day 1 n=7,0 | 9.5 (31.71) |
  Alopecia CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Alopecia CFB at Cycle 13, Day 1 n=5,0 | 13.3 (29.81) |
  Alopecia CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Alopecia CFB at Cycle 15, Day 1 n=5,0 | 0.0 (0.00) |
  Alopecia CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Alopecia CFB at Cycle 17, Day 1 n=4,0 | 0.0 (0.00) |
  Alopecia CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Alopecia CFB at Cycle 19, Day 1 n=5,0 | 20.0 (29.81) |
  Alopecia CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Alopecia CFB at Cycle 21, Day 1 n=4,0 | 8.3 (16.67) |
  Alopecia CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Alopecia CFB at Cycle 23, Day 1 n=2,0 | 16.7 (23.57) |
  Alopecia CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Alopecia CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Alopecia CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Alopecia CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Alopecia CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Alopecia CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Pain in Chest CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Pain in Chest CFB at Cycle 3, Day 1 n=12,4 | -19.4 (22.29) | -8.3 (41.94)
  Pain in Chest CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Pain in Chest CFB at Cycle 5, Day 1 n=8,3 | -8.3 (29.55) | -11.1 (50.92)
  Pain in Chest CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Pain in Chest CFB at Cycle 7, Day 1 n=8,1 | -25.0 (15.43) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Pain in Chest CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Pain in Chest CFB at Cycle 9, Day 1 n=7,2 | -23.8 (25.20) | 0.0 (47.14)
  Pain in Chest CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Pain in Chest CFB at Cycle 11, Day 1 n=7,0 | -4.8 (23.00) |
  Pain in Chest CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Chest CFB at Cycle 13, Day 1 n=5,0 | -13.3 (18.26) |
  Pain in Chest CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Chest CFB at Cycle 15, Day 1 n=5,0 | -13.3 (18.26) |
  Pain in Chest CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain in Chest CFB at Cycle 17, Day 1 n=4,0 | 0.0 (27.22) |
  Pain in Chest CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Chest CFB at Cycle 19, Day 1 n=5,0 | -20.0 (18.26) |
  Pain in Chest CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain in Chest CFB at Cycle 21, Day 1 n=4,0 | 0.0 (38.49) |
  Pain in Chest CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Chest CFB at Cycle 23, Day 1 n=2,0 | 33.3 (47.14) |
  Pain in Chest CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Chest CFB at Cycle 25, Day 1 n=2,0 | 16.7 (23.57) |
  Pain in Chest CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Chest CFB at Cycle 27, Day 1 n=2,0 | 16.7 (23.57) |
  Pain in Chest CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Chest CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Pain in Arm or Shoulder CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Pain in Arm or Shoulder CFB at Cycle 3, Day 1 n=12,4 | -2.8 (30.01) | -33.3 (38.49)
  Pain in Arm or Shoulder CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Pain in Arm or Shoulder CFB at Cycle 5, Day 1 n=8,3 | -8.3 (15.43) | -22.2 (19.25)
  Pain in Arm or Shoulder CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Pain in Arm or Shoulder CFB at Cycle 7, Day 1 n=8,1 | -8.3 (34.50) | -33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Pain in Arm or Shoulder CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Pain in Arm or Shoulder CFB at Cycle 9, Day 1 n=7,2 | -9.5 (37.09) | -16.7 (70.71)
  Pain in Arm or Shoulder CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Pain in Arm or Shoulder CFB at Cycle 11, Day 1 n=7,0 | -9.5 (53.45) |
  Pain in Arm or Shoulder CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Arm or Shoulder CFB at Cycle 13, Day 1 n=5,0 | -6.7 (36.51) |
  Pain in Arm or Shoulder CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Arm or Shoulder CFB at Cycle 15, Day 1 n=5,0 | -26.7 (49.44) |
  Pain in Arm or Shoulder CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain in Arm or Shoulder CFB at Cycle 17, Day 1 n=4,0 | -16.7 (57.74) |
  Pain in Arm or Shoulder CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Arm or Shoulder CFB at Cycle 19, Day 1 n=5,0 | -6.7 (59.63) |
  Pain in Arm or Shoulder CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain in Arm or Shoulder CFB at Cycle 21, Day 1 n=4,0 | -25.0 (56.93) |
  Pain in Arm or Shoulder CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Arm or Shoulder CFB at Cycle 23, Day 1 n=2,0 | -16.7 (23.57) |
  Pain in Arm or Shoulder CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Arm or Shoulder CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Pain in Arm or Shoulder CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Arm or Shoulder CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Pain in Arm or Shoulder CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Arm or Shoulder CFB at Cycle 29, Day 1 n=2,0 | -50.0 (70.71) |
  Pain in Other Parts CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Pain in Other Parts CFB at Cycle 3, Day 1 n=12,4 | -8.3 (37.94) | -8.3 (16.67)
  Pain in Other Parts CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Pain in Other Parts CFB at Cycle 5, Day 1 n=8,3 | -12.5 (17.25) | 0.0 (0.00)
  Pain in Other Parts CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Pain in Other Parts CFB at Cycle 7, Day 1 n=8,1 | -12.5 (35.36) | 33.3 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Pain in Other Parts CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Pain in Other Parts CFB at Cycle 9, Day 1 n=7,2 | -9.5 (16.27) | 16.7 (23.57)
  Pain in Other Parts CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Pain in Other Parts CFB at Cycle 11, Day 1 n=7,0 | 4.8 (35.63) |
  Pain in Other Parts CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Other Parts CFB at Cycle 13, Day 1 n=5,0 | -6.7 (14.91) |
  Pain in Other Parts at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Other Parts at Cycle 15, Day 1 n=5,0 | -13.3 (18.26) |
  Pain in Other Parts CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain in Other Parts CFB at Cycle 17, Day 1 n=4,0 | 16.7 (43.03) |
  Pain in Other Parts CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain in Other Parts CFB at Cycle 19, Day 1 n=5,0 | 20.0 (44.72) |
  Pain in Other Parts CFB at Cycle 21, Day 1 n=: number analyzed (Participants) | 4 | 0
  Pain in Other Parts CFB at Cycle 21, Day 1 n= | 8.3 (16.67) |
  Pain in Other Parts CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Other Parts CFB at Cycle 23, Day 1 n=2,0 | 0.0 (0.00) |
  Pain in Other Parts CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Other Parts CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Pain in Other Parts CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Other Parts CFB at Cycle 27, Day 1 n=2,0 | -16.7 (23.57) |
  Pain in Other Parts CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain in Other Parts CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |

19. Secondary Outcome: Change From Baseline in Score as Per European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L is a standardized measure to assess the overall health-related quality of life in patients. The EQ-5D-5L consists of 2 parts- the descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with 5 levels: from 1 (no problems) to 5 (extreme problems). The EQ VAS is a self-perceived health score assessed using a visual analogue scale that ranges from 0 (the worst imaginable health) to 100 (the best imaginable health), with higher scores indicating higher health utility. CFB = change from baseline.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
score on a scale
  Anxiety/Depression CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Anxiety/Depression CFB at Cycle 3, Day 1 n=12,4 | -0.6 (0.79) | 0.0 (0.82)
  Anxiety/Depression CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Anxiety/Depression CFB at Cycle 5, Day 1 n=8,3 | -0.3 (1.16) | -0.7 (1.53)
  Anxiety/Depression CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Anxiety/Depression CFB at Cycle 7, Day 1 n=8,1 | -0.3 (1.39) | -1.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Anxiety/Depression CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Anxiety/Depression CFB at Cycle 9, Day 1 n=7,2 | 0.0 (1.41) | 0.0 (1.41)
  Anxiety/Depression CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Anxiety/Depression CFB at Cycle 11, Day 1 n=7,0 | 0.4 (0.98) |
  Anxiety/Depression CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Anxiety/Depression CFB at Cycle 13, Day 1 n=5,0 | -0.4 (1.14) |
  Anxiety/Depression CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Anxiety/Depression CFB at Cycle 15, Day 1 n=5,0 | -0.2 (1.10) |
  Anxiety/Depression CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Anxiety/Depression CFB at Cycle 17, Day 1 n=4,0 | 0.5 (1.29) |
  Anxiety/Depression CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Anxiety/Depression CFB at Cycle 19, Day 1 n=5,0 | -0.2 (0.84) |
  Anxiety/Depression CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Anxiety/Depression CFB at Cycle 21, Day 1 n=4,0 | 0.5 (1.73) |
  Anxiety/Depression CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Anxiety/Depression CFB at Cycle 23, Day 1 n=2,0 | 0.0 (0.00) |
  Anxiety/Depression CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Anxiety/Depression CFB at Cycle 25, Day 1 n=2,0 | -0.5 (0.71) |
  Anxiety/Depression CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Anxiety/Depression CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Anxiety/Depression CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Anxiety/Depression CFB at Cycle 29, Day 1 n=2,0 | 0.5 (2.12) |
  EQ VAS Score CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  EQ VAS Score CFB at Cycle 3, Day 1 n=12,4 | 11.7 (17.99) | 10.3 (11.32)
  EQ VAS Score CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  EQ VAS Score CFB at Cycle 5, Day 1 n=8,3 | 12.6 (12.47) | 10.3 (5.03)
  EQ VAS Score CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  EQ VAS Score CFB at Cycle 7, Day 1 n=8,1 | 7.6 (15.34) | -6.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  EQ VAS Score CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  EQ VAS Score CFB at Cycle 9, Day 1 n=7,2 | 6.7 (18.29) | 5.0 (8.49)
  EQ VAS Score CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  EQ VAS Score CFB at Cycle 11, Day 1 n=7,0 | -1.4 (14.36) |
  EQ VAS Score CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  EQ VAS Score CFB at Cycle 13, Day 1 n=5,0 | 10.8 (21.23) |
  EQ VAS Score CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  EQ VAS Score CFB at Cycle 15, Day 1 n=5,0 | 1.6 (10.88) |
  EQ VAS Score CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  EQ VAS Score CFB at Cycle 17, Day 1 n=4,0 | -4.5 (13.77) |
  EQ VAS Score CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  EQ VAS Score CFB at Cycle 19, Day 1 n=5,0 | 2.0 (12.27) |
  EQ VAS Score CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  EQ VAS Score CFB at Cycle 21, Day 1 n=4,0 | -5.0 (10.80) |
  EQ VAS Score CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  EQ VAS Score CFB at Cycle 23, Day 1 n=2,0 | -7.5 (17.68) |
  EQ VAS Score CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  EQ VAS Score CFB at Cycle 25, Day 1 n=2,0 | -4.0 (26.87) |
  EQ VAS Score CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  EQ VAS Score CFB at Cycle 27, Day 1 n=2,0 | -17.0 (16.97) |
  EQ VAS Score CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  EQ VAS Score CFB at Cycle 29, Day 1 n=2,0 | -16.5 (9.19) |
  Pain/Discomfort CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Pain/Discomfort CFB at Cycle 3, Day 1 n=12,4 | -0.3 (0.89) | 0.3 (0.96)
  Pain/Discomfort CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Pain/Discomfort CFB at Cycle 5, Day 1 n=8,3 | 0.1 (0.99) | 0.0 (1.00)
  Pain/Discomfort CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Pain/Discomfort CFB at Cycle 7, Day 1 n=8,1 | 0.4 (1.06) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Pain/Discomfort CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Pain/Discomfort CFB at Cycle 9, Day 1 n=7,2 | 0.0 (0.82) | 1.0 (0.00)
  Pain/Discomfort CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Pain/Discomfort CFB at Cycle 11, Day 1 n=7,0 | 0.1 (1.57) |
  Pain/Discomfort CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain/Discomfort CFB at Cycle 13, Day 1 n=5,0 | 0.6 (1.52) |
  Pain/Discomfort CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain/Discomfort CFB at Cycle 15, Day 1 n=5,0 | 0.0 (1.58) |
  Pain/Discomfort CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain/Discomfort CFB at Cycle 17, Day 1 n=4,0 | 0.8 (2.22) |
  Pain/Discomfort CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Pain/Discomfort CFB at Cycle 19, Day 1 n=5,0 | -0.2 (1.48) |
  Pain/Discomfort CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Pain/Discomfort CFB at Cycle 21, Day 1 n=4,0 | 0.3 (1.71) |
  Pain/Discomfort CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain/Discomfort CFB at Cycle 23, Day 1 n=2,0 | 2.0 (0.00) |
  Pain/Discomfort CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain/Discomfort CFB at Cycle 25, Day 1 n=2,0 | 1.0 (1.41) |
  Pain/Discomfort CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain/Discomfort CFB at Cycle 27, Day 1 n=2,0 | 1.5 (0.71) |
  Pain/Discomfort CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Pain/Discomfort CFB at Cycle 29, Day 1 n=2,0 | 0.5 (0.71) |
  Mobility CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Mobility CFB at Cycle 3, Day 1 n=12,4 | -0.3 (0.75) | -0.3 (0.96)
  Mobility CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Mobility CFB at Cycle 5, Day 1 n=8,3 | -0.4 (0.92) | 0.7 (1.53)
  Mobility CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Mobility CFB at Cycle 7, Day 1 n=8,1 | -0.1 (0.83) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Mobility CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Mobility CFB at Cycle 9, Day 1 n=7,2 | -0.4 (0.98) | 1.0 (1.41)
  Mobility CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Mobility CFB at Cycle 11, Day 1 n=7,0 | -0.1 (1.07) |
  Mobility CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Mobility CFB at Cycle 13, Day 1 n=5,0 | -0.2 (0.84) |
  Mobility CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Mobility CFB at Cycle 15, Day 1 n=5,0 | 0.2 (0.45) |
  Mobility CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Mobility CFB at Cycle 17, Day 1 n=4,0 | 0.3 (0.96) |
  Mobility CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Mobility CFB at Cycle 19, Day 1 n=5,0 | 0.0 (1.00) |
  Mobility CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Mobility CFB at Cycle 21, Day 1 n=4,0 | -0.3 (0.96) |
  Mobility CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Mobility CFB at Cycle 23, Day 1 n=2,0 | 0.5 (0.71) |
  Mobility CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Mobility CFB at Cycle 25, Day 1 n=2,0 | 0.5 (0.71) |
  Mobility CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Mobility CFB at Cycle 27, Day 1 n=2,0 | 1.0 (1.41) |
  Mobility CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Mobility CFB at Cycle 29, Day 1 n=2,0 | 0.0 (0.00) |
  Self-Care CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Self-Care CFB at Cycle 3, Day 1 n=12,4 | -0.2 (0.72) | 0.0 (0.00)
  Self-Care CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Self-Care CFB at Cycle 5, Day 1 n=8,3 | 0.5 (0.76) | 0.0 (0.00)
  Self-Care CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Self-Care CFB at Cycle 7, Day 1 n=8,1 | 0.0 (1.20) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Self-Care CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Self-Care CFB at Cycle 9, Day 1 n=7,2 | 0.1 (1.35) | 0.0 (0.00)
  Self-Care CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Self-Care CFB at Cycle 11, Day 1 n=7,0 | 0.1 (1.46) |
  Self-Care CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Self-Care CFB at Cycle 13, Day 1 n=5,0 | 0.0 (1.22) |
  Self-Care CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Self-Care CFB at Cycle 15, Day 1 n=5,0 | 0.0 (1.22) |
  Self-Care CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Self-Care CFB at Cycle 17, Day 1 n=4,0 | 0.0 (1.63) |
  Self-Care CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Self-Care CFB at Cycle 19, Day 1 n=5,0 | 0.0 (1.58) |
  Self-Care CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Self-Care CFB at Cycle 21, Day 1 n=4,0 | -0.3 (1.71) |
  Self-Care CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Self-Care CFB at Cycle 23, Day 1 n=2,0 | 1.0 (1.41) |
  Self-Care CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Self-Care CFB at Cycle 25, Day 1 n=2,0 | 1.0 (1.41) |
  Self-Care CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Self-Care CFB at Cycle 27, Day 1 n=2,0 | 1.0 (1.41) |
  Self-Care CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Self-Care CFB at Cycle 29, Day 1 n=2,0 | -0.5 (0.71) |
  Usual Activities CFB at Cycle 3, Day 1 n=12,4: number analyzed (Participants) | 12 | 4
  Usual Activities CFB at Cycle 3, Day 1 n=12,4 | -0.7 (1.23) | 1.3 (0.50)
  Usual Activities CFB at Cycle 5, Day 1 n=8,3: number analyzed (Participants) | 8 | 3
  Usual Activities CFB at Cycle 5, Day 1 n=8,3 | -0.9 (1.55) | 0.7 (0.58)
  Usual Activities CFB at Cycle 7, Day 1 n=8,1: number analyzed (Participants) | 8 | 1
  Usual Activities CFB at Cycle 7, Day 1 n=8,1 | -0.8 (1.28) | 0.0 (NA) — Standard deviation was not calculable due the single data point for the mean value.
  Usual Activities CFB at Cycle 9, Day 1 n=7,2: number analyzed (Participants) | 7 | 2
  Usual Activities CFB at Cycle 9, Day 1 n=7,2 | -0.7 (0.95) | 1.5 (0.71)
  Usual Activities CFB at Cycle 11, Day 1 n=7,0: number analyzed (Participants) | 7 | 0
  Usual Activities CFB at Cycle 11, Day 1 n=7,0 | -0.7 (1.38) |
  Usual Activities CFB at Cycle 13, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Usual Activities CFB at Cycle 13, Day 1 n=5,0 | -0.8 (0.84) |
  Usual Activities CFB at Cycle 15, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Usual Activities CFB at Cycle 15, Day 1 n=5,0 | -0.4 (0.55) |
  Usual Activities CFB at Cycle 17, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Usual Activities CFB at Cycle 17, Day 1 n=4,0 | -0.3 (0.50) |
  Usual Activities CFB at Cycle 19, Day 1 n=5,0: number analyzed (Participants) | 5 | 0
  Usual Activities CFB at Cycle 19, Day 1 n=5,0 | -0.4 (0.55) |
  Usual Activities CFB at Cycle 21, Day 1 n=4,0: number analyzed (Participants) | 4 | 0
  Usual Activities CFB at Cycle 21, Day 1 n=4,0 | -0.8 (0.96) |
  Usual Activities CFB at Cycle 23, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Usual Activities CFB at Cycle 23, Day 1 n=2,0 | 0.5 (0.71) |
  Usual Activities CFB at Cycle 25, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Usual Activities CFB at Cycle 25, Day 1 n=2,0 | 0.0 (0.00) |
  Usual Activities CFB at Cycle 27, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Usual Activities CFB at Cycle 27, Day 1 n=2,0 | 0.0 (0.00) |
  Usual Activities CFB at Cycle 29, Day 1 n=2,0: number analyzed (Participants) | 2 | 0
  Usual Activities CFB at Cycle 29, Day 1 n=2,0 | 1.0 (1.41) |

20. Secondary Outcome: Time to Symptom Deterioration for Chest Pain, Cough and Dyspnea Assessed Using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Lung Cancer Module (QLQ-LC13)
Description: EORTC QLQ-LC13 is a 13-item lung cancer specific questionnaire. The assessments here included chest pain, cough, and dyspnea and were based on their presence over the previous week. All but the pain domain were scored on a 4 point Likert scale ranging from "not at all" to "very much." Pain was scored based on its presence, yes or no. Scores were averaged and transformed to 0 to 100. A higher score indicated a higher presence of symptoms. Time to symptom deterioration for chest pain, cough and dyspnea was assessed. Deterioration was assessed by the investigator.
Time Frame: Cycle (C) 1 Day (D) 1, C3 D1 and then every 6 weeks up to approximately 21 months, end of treatment and 6, 12, 18 weeks post treatment. Each cycle duration was 21 days.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
months
  Coughing | 13.9 [2.76 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 2.9 [1.38 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
  Dyspnea | 5.7 [2.76 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 2.9 [1.38 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.
  Pain in chest | 11.1 [2.76 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 2.9 [1.45 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

21. Secondary Outcome: Time to Deterioration for Global Health Status /QoL Assessed Using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. The questionnaire is composed of both multi-item scales and single-item measures based on the participants experience over the past week. These include five domains (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/HRQoL scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Time to deterioration in QoL from EORTC-QLQ-C30 was assessed. Deterioration was assessed by the investigator.
Time Frame: as for outcome 20
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 7
months | NA [2.92 to NA] — The median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [1.38 to NA] — The median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

22. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths due to any cause were collected from first dose of study medication to 30 days after the last dose of study treatment. Post-treatment survival follow-up deaths were collected from Day 31 after last dose of study medication to the data cut-off date.
Time Frame: On-treatment deaths: Up to approximately 117 weeks. Post-treatment survival follow-up deaths: Up to an additional 36 weeks.
Population: The safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Capmatinib | Docetaxel
Number analyzed (Participants) | 15 | 6
Participants
  On-treatment deaths | 2 | 0
  Post-treatment deaths | 7 | 5
  All deaths | 9 | 5

ADVERSE EVENTS:
Time Frame: From day of first dose of study medication to last dose of study medication plus 30 days, up to approximately 117 weeks. Deaths were collected in the post-treatment phase from 31 days after last dose of study medication until the end of the study, up to approximately 36 additional weeks. These were not considered AEs.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival includes participants who entered the post-treatment survival follow-up period.
Groups:
- Capmatinib (On-treatment): 400 mg, capmatinib tablets, administered orally twice daily
- Docetaxel (On-treatment): Docetaxel 75 mg/m^2 solution administered by intravenous infusion on Day 1 of every 21-day cycle
- Capmatinib Extension Crossover Treatment (On-treatment): 400 mg, capmatinib tablets, administered orally twice daily to participants treated with docetaxel who crossed over to capmatinib treatment.
- Capmatinib (Post-treatment Survival Follow-up); Docetaxel (Post-treatment Survival Follow-up): Deaths collected in the post-treatment survival follow-up period (starting from Day 31 post-treatment). No AEs were collected during this period.
Arm/Group | Capmatinib (On-treatment) | Docetaxel (On-treatment) | Capmatinib Extension Crossover Treatment (On-treatment) | Capmatinib (Post-treatment Survival Follow-up) | Docetaxel (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 2/15 | 0/6 | 0/5 | 7/13 | 5/6
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/6 | 1/5 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 14/15 | 5/6 | 4/5 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capmatinib (On-treatment) (N=15) | Docetaxel (On-treatment) (N=6) | Capmatinib Extension Crossover Treatment (On-treatment) (N=5) | Capmatinib (Post-treatment Survival Follow-up) (N=0) | Docetaxel (Post-treatment Survival Follow-up) (N=0)
Chest pain (General disorders) | 0 | 1 | 1 | NA | NA
Pain (General disorders) | 1 | 0 | 0 | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | NA | NA
Sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capmatinib (On-treatment) (N=15) | Docetaxel (On-treatment) (N=6) | Capmatinib Extension Crossover Treatment (On-treatment) (N=5) | Capmatinib (Post-treatment Survival Follow-up) (N=0) | Docetaxel (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | NA | NA
Palpitations (Cardiac disorders) | 1 | 0 | 0 | NA | NA
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | NA | NA
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | NA | NA
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | NA | NA
Deafness (Ear and labyrinth disorders) | 2 | 0 | 0 | NA | NA
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 1 | NA | NA
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | NA | NA
Myxoedema (Endocrine disorders) | 1 | 0 | 0 | NA | NA
Eye pruritus (Eye disorders) | 1 | 0 | 0 | NA | NA
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | NA | NA
Lacrimation increased (Eye disorders) | 1 | 2 | 2 | NA | NA
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Constipation (Gastrointestinal disorders) | 4 | 1 | 1 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | NA | NA
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 5 | 1 | 1 | NA | NA
Odynophagia (Gastrointestinal disorders) | 3 | 0 | 0 | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | NA | NA
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 6 | 0 | 0 | NA | NA
Asthenia (General disorders) | 4 | 2 | 2 | NA | NA
Fatigue (General disorders) | 1 | 1 | 1 | NA | NA
Gait disturbance (General disorders) | 1 | 0 | 0 | NA | NA
Mucosal inflammation (General disorders) | 1 | 0 | 0 | NA | NA
Oedema (General disorders) | 2 | 0 | 0 | NA | NA
Oedema peripheral (General disorders) | 10 | 0 | 0 | NA | NA
Peripheral swelling (General disorders) | 1 | 0 | 0 | NA | NA
Pyrexia (General disorders) | 3 | 0 | 0 | NA | NA
Suprapubic pain (General disorders) | 1 | 0 | 0 | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA
Bronchitis (Infections and infestations) | 1 | 0 | 0 | NA | NA
COVID-19 (Infections and infestations) | 1 | 0 | 0 | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 2 | 2 | NA | NA
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | NA | NA
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | NA | NA
Influenza (Infections and infestations) | 0 | 1 | 1 | NA | NA
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | NA | NA
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | NA | NA
Rhinolaryngitis (Infections and infestations) | 0 | 1 | 1 | NA | NA
Sinusitis (Infections and infestations) | 0 | 1 | 1 | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | NA | NA
Amylase increased (Investigations) | 2 | 0 | 0 | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | NA | NA
Blood albumin decreased (Investigations) | 1 | 0 | 0 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | NA | NA
Blood cholesterol increased (Investigations) | 0 | 1 | 1 | NA | NA
Blood creatinine increased (Investigations) | 4 | 0 | 0 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | NA | NA
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0 | NA | NA
Creatinine renal clearance increased (Investigations) | 1 | 0 | 0 | NA | NA
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | NA | NA
Lipase increased (Investigations) | 1 | 0 | 0 | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | NA | NA
Protein total decreased (Investigations) | 1 | 0 | 0 | NA | NA
Transaminases increased (Investigations) | 1 | 0 | 0 | NA | NA
Weight decreased (Investigations) | 1 | 0 | 0 | NA | NA
Weight increased (Investigations) | 3 | 0 | 0 | NA | NA
White blood cell count decreased (Investigations) | 0 | 1 | 1 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 1 | NA | NA
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | NA | NA
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA
Dizziness (Nervous system disorders) | 3 | 0 | 0 | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 1 | 1 | NA | NA
Headache (Nervous system disorders) | 1 | 0 | 0 | NA | NA
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | NA | NA
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | NA | NA
Somnolence (Nervous system disorders) | 1 | 0 | 0 | NA | NA
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | NA | NA
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | NA | NA
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | NA | NA
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA
Penile dermatitis (Reproductive system and breast disorders) | 0 | 1 | 1 | NA | NA
Perineal rash (Reproductive system and breast disorders) | 0 | 1 | 1 | NA | NA
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | NA | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 4 | NA | NA
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | NA | NA
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | NA | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | NA | NA
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | NA | NA
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | NA | NA
Embolism (Vascular disorders) | 0 | 1 | 1 | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | 0 | NA | NA
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04427072/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04427072/SAP_001.pdf